CLINICAL TRIAL: NCT02962141
Title: Evaluation of the Safety and Efficacy of the Paclitaxel Eluting Hemodialysis Shunt Balloon Dilatation Catheter (APERTO) in Treatment of Hemodialysis Arteriovenous Fistulae Stenosis: A Prospective, Multicenter, Randomized, Controlled Clinical Study
Brief Title: A Study of Hemodialysis Arteriovenous Fistulae Stenosis Treated With APERTO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ZhuHai Cardionovum Medical Device Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APERTO-2015-01
Record Dates: First submitted 2016-11-08; First posted 2016-11-11 (Estimated); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Peripheral Arterial Disease; Fistula
Keywords: drug eluting balloon, Arteriovenous Fistulae
MeSH Terms: conditions — Peripheral Arterial Disease; Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- APERTO OTW group (Experimental): in the APERTO OTW group the subject will be treated with APERTO OTW balloon (Paclitaxel Releasing Peripheral Balloon Dilatation Catheter)
  Interventions: Device: Paclitaxel Releasing Peripheral Balloon Dilatation Catheter
- OHICHO II group (Active Comparator): in the OHICHO II group the subject will be treated with OHICHO II balloon (Balloon Dilatation Catheter)
  Interventions: Device: Balloon Dilatation Catheter

INTERVENTIONS:
Device: Paclitaxel Releasing Peripheral Balloon Dilatation Catheter — Treatment group
  Other Names: APERTO OTW
  Arms: APERTO OTW group
Device: Balloon Dilatation Catheter — Control group
  Other Names: OHICHO II
  Arms: OHICHO II group

SUMMARY:
To evaluate the safety and efficacy of Paclitaxel Eluting Hemodialysis Shunt Balloon Dilatation Catheter (APERTO) compared with the Balloon Dilatation catheter (OHICHO II) for the treatment of Arteriovenous Fistulae Stenosis in patients undergoing hemodialysis.

DETAILED DESCRIPTION:
To evaluate the safety and efficacy of the Paclitaxel Eluting Hemodialysis Shunt Balloon Dilatation Catheter (APERTO) compared with the Balloon Dilatation catheter (OHICHO II) for the treatment of Arteriovenous Fistulae Stenosis in patients undergoing hemodialysis.

This is a prospective, multi-center, randomized controlled, open-label, superiority study. A total of 160 subjects will be enrolled from 10 sites in China. All subjects enrolled will be randomly assigned to the test group (APERTO group, n=80) and the control group (OHICHO II group, n=80) with randomized allocation ratio of 1:1. Subjects in the test group and the control group will be treated with APERTO OTW or OHICHO II respectively.

ELIGIBILITY:
Inclusion criteria:

Patients must meet all of the following criteria:

* Age ≥ 18 years and ≤ 75 years, male or female.
* Patient or legally authorized representative can understand the purpose of this clinic trial. He or She volunteers to participate in this trial and can provide written informed consent, and is willing to accept the scheduled follow-up in specific time points.
* Angiography, ultrasound or clinical diagnosis shows that patients have hemodialysis access dysfunction due to stenosis lesions.
* Patients with indications of the percutaneous endovascular therapy, that is, the AVF stenosis is related to hemodynamics and ≥ 50%, and with any of the following clinical and physiological abnormalities (referred to NKF-K/DOQI guideline definitions):

  1. Thrombosis in the AVF;
  2. Elevated venous pressure during dialysis
  3. Obvious abnormality in recirculation measurements
  4. Abnormal physical examination findings
  5. Unexplained decreases in dialysis dose
  6. Decreased access flow
* Target lesion is a de novo or restenosis. The number of target lesions is 1.
* Target lesion consists of a single lesion or a multiple lesions with target lesion length ≤ 40 mm.
* Target lesion(s) is located in the reflux vein which is from the anastomosis of native arteriovenous fistula (AVF) to the distal end of subclavian vein, except the anastomosis of native AVF.
* If patient has non-target lesion, it must be successfully treated using PTA before treating target lesion.
* Reference vessel diameter of target lesion ≥ 4.0 mm and ≤ 7.0 mm by visual estimate (determined by angiography or DUS).
* Hemodialysis access previously used (mature AVF) can no longer be successfully used due to insufficient shunt flow volume caused by local lumen stenosis.

Exclusion criteria:

Patients will be excluded if any of the following conditions applies:

* Patients who have participated in another investigational drug or device trial.
* Patients who have been enrolled in this trial previously.
* Women of childbearing age with negative pregnancy test before procedure, and breastfeeding women.
* Any major surgical procedure (such as thoracotomy, craniotomy, etc.) within 30 days prior to the procedure.
* Any planned major surgical procedure (such as thoracotomy, craniotomy, etc.) within 30 days of entry into this study
* Immature AVF, which cannot be used for Dialysis or has not been used successfully due to insufficient lumen diameter to ensure successfully puncture and insufficient shunt flow volume.
* Patients with AVG.
* AVF has been previously implanted with stent.
* Lesion in AVF has been previously treated with DEB.
* Target lesion is located in the anastomosis of native AVF.
* Known allergies or intolerance to Paclitaxel or contrast medium.
* Life expectancy < 1 year
* Patients with comitans systemic lupus erythematosus and ANCA associated vasculitis.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2016-10; Primary Completion 2018-01 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Primary patency rate of the target lesion | at 6 month post procedure
  Primary patency is defined as freedom from restenosis as determined by DUS Peak Systolic Velocity Ratio (PSVR) ≤ 2.0 and freedom from clinically-driven target lesion revascularization (CD-TLR).
  Restenosis is defined as PSVR> 2.0 determined by independent DUS laboratory. Clinically-driven target lesion revascularization (CD-TLR) is defined as any re-intervention in target lesion (+/-5mm proximal or distal of the target lesion) determined by DUS due to clinical symptoms or dialysis indicators showing that it is unable to perform dialysis.

SECONDARY OUTCOMES:
Device Success | intraoperative
  Device Success is defined as ability of the Device to be delivered, inflated at pressure ≤ RBP, and retrieved from the Target Lesion without burst.
Technical Success | intraoperative
  Technical Success is defined as the residual stenosis of the lumen diameter ≤ 30% after treatment with either APERTO OTW or OHICHO II (compared with the referred vessel diameter of the nearest veins with no aneurysm).
Clinical Success | at 1 month
  Clinical Success is defined as improvement in hemodialysis access function and resumption of normal dialysis for at least one dialysis session after the index procedure.
Procedural Success | at 1 month
  Procedural Success is defined as technical success without the occurrence of MAE during the hospitalization or day of treatment (MAE defined here as: death, stroke, thrombotic occlusion, allergic reaction, pulmonary events (including pulmonary edema)
MAE rates (death or stroke) | at 1 month, 3 months, 6 months, and 12 months post procedure.
The diameter stenosis rate in target lesion | at 6 months post procedure
  The diameter stenosis (%)=100% × (1-(MLD/RVD))
Clinical-driven Target Lesion Revascularization (CD-TLR) | in1st, 3rd, 6th, 12th month post operation
  CD-TLR is defined as any re-intervention in target lesion (+/-5mm proximal or distal of the target lesion) determined by DUS due to clinical symptoms or dialysis indicators showing that it is unable to perform dialysis.
Clinical-driven Target Shunt Revascularization (CD-TSR) | in 1st, 3rd, 6th, 12th month post operation
  Target Shunt is defined as the reflux vein, which is from the anastomotic stoma of native arteriovenous fistula (AVF) to the distal end of the subclavian vein.
  CD-TSR is defined as any re-intervention in target lesion due to clinical symptoms or inability to perform dialysis.

CONTACTS AND LOCATIONS:
Overall Officials: Qizhuang Jin, professor, Principal Investigator — Peking University First Hospital
Locations (9):
- China (9):
  - Hainan General Hospital, Haikou, Hainan
  - The First Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Sir Run Run Shaw Hospital School of Medicine, Zhejiang University, Hangzhou, Zhejiang
  - The First Hospital of Zhejiang Province, Hangzhou, Zhejiang
  - Beijing Tongren Hospital, Capital Medical University, Beijing
  - Longhua Hospital Shanghai University of Tranditional Chinese Medicine, Shanghai

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Yin Y, Shi Y, Cui T, Li H, Chen J, Zhang L, Yu Z, Li H, Yan Y, Wu K, Jin Q. Efficacy and Safety of Paclitaxel-Coated Balloon Angioplasty for Dysfunctional Arteriovenous Fistulas: A Multicenter Randomized Controlled Trial. Am J Kidney Dis. 2021 Jul;78(1):19-27.e1. doi: 10.1053/j.ajkd.2020.11.022. Epub 2021 Jan 5. PMID 33418016